CLINICAL TRIAL: NCT00953719
Title: Delta Ceramax 36 mm Ceramic-on-Ceramic Acetabular Cup Prosthesis Study
Brief Title: 36 mm Ceramic-on-Ceramic Acetabular Cup Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COC 36 mm
Record Dates: First submitted 2009-06-03; First posted 2009-08-06 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Non-inflammatory Degenerative Joint Disease
Keywords: Hip arthroplasty; Acetabular cup; Ceramic-on-polyethylene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 36 mm (Active Comparator): 36 mm ceramic head on ceramic acetabular liner
  Interventions: Device: 36 mm ceramic head on a ceramic acetabular liner
- 28 mm ceramic-on-polyethylene (Other): 28 mm ceramic-on-polyethylene historical control
  Interventions: Device: 28 mm ceramic head on a polyethylene acetabular liner

INTERVENTIONS:
Device: 36 mm ceramic head on a ceramic acetabular liner — Total hip replacement with a 36 mm ceramic head on a ceramic liner
  Other Names: Delta Ceramax head on a ceramic liner.
  Arms: 36 mm
Device: 28 mm ceramic head on a polyethylene acetabular liner — Total hip replacement with a 28 mm ceramic head on a polyethylene liner.
  Other Names: Delta Ceramax head on a polyethylene liner
  Arms: 28 mm ceramic-on-polyethylene

SUMMARY:
This study is a supplement to the 28 mm Ceramic-on-Ceramic study which was designed to evaluate artificial hips with a 28 mm ceramic head and liner to determine whether they perform as well as artificial hips with a 28 mm ceramic head and a polyethylene liner.

This arm of the study is designed to compare a 36 mm ceramic head and sleeve with a subset of the control (28mm ceramic head and a polyethylene sleeve) from the original study (G030075) (NCT#00208507) with additional follow-up, to determine if they perform as well.

DETAILED DESCRIPTION:
Total Hip Arthroplasty (THA) is the surgical reconstruction of the hip joint through replacement of the femoral head and the acetabular articulating surfaces with fixed prosthetic devices. The goals of THA are relief from pain, restoration of function, and correction of deformity. THA is one of the most common adult reconstructive procedures. Over the past 25 years, patients who have needed to have their hip joint replaced, either due to trauma or arthritic disease, typically have had their hip joint bone articular surfaces replaced with a metal hip stem, metal ball head (either stainless steel or chrome cobalt) and a plastic acetabular cup (metal/metal/plastic). While the basic device has remained essentially unchanged over that period, technological advancements in implant designs and materials, and improvements in surgical technique and instrumentation have made THA one of the most durable and successful procedures in medicine. Reproducible, high-quality, short-term and mid-term results are attained regularly, and total hip replacements commonly last 10 to 15 years and longer. The success of this procedure has allowed its expansion into a wider, and often younger and more active population.

In spite of the improvements in THA, little change has occurred for the acetabular cup liner, which is usually made out of Ultra High Molecular Weight Polyethylene plastic (UHMWPe). Because it is plastic and inherently soft and somewhat pliable under load, the cup's articular surface must inevitability wear and produce debris. This biologic response is now thought to be a significant contributor to prosthetic component loosening, a primary failure mode of THR. UHMWPe also degrades with time in the body. As concerns about polyethylene wear and the associated untoward effects of the generated wear debris, and as THA continues to be used in younger and higher-demand patients with increasing life expectancies, interest in ceramic on ceramic total hip prosthesis has been renewed.

An alumina ceramic-on-ceramic acetabular coupling has been employed as an alternative to metal/polyethylene couplings. This ceramic-on-ceramic coupling has many advantages, including the elimination of polyethylene from the device system, wear rates that are appreciably less than those experienced with metal/polyethylene couplings and reduced biologic reactivity. The potential benefits of an alumina ceramic/ceramic bearing are significant.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease. Composite diagnoses of NIDJD include osteoarthritis, avascular necrosis, post-traumatic arthritis, slipped capital femoral epiphysis (SCFE), fracture of the pelvis, and developmental dysplasia.
* X-ray evaluation confirms the presence of NIDJD
* Femoral and acetabular bone stock is sufficient, regarding strength and shape, and is suitable to receive the implants.
* Individuals 20 to 75 years of age at the time of surgery
* Patients with a previous total hip replacement of the contralateral leg who have a pain rating of none or slight and who are at least one year post arthroplasty are eligible for participation in the study.
* Harris Hip Score of 70 or lower
* Pain at least Moderate

Exclusion Criteria:

* Presence of a previous prosthetic hip replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) in the hip joint to be operated.
* Previous Girdlestone procedure (resection arthroplasty) or surgical fusion of the hip to be operated.
* Acute femoral neck fracture.
* Above knee amputation of the contralateral and/or ipsilateral leg.
* Patients with bilateral degenerative joint disease requiring staged or simultaneous hip replacements.
* Patients with an existing total hip arthroplasty in the contralateral hip with a Harris Hip pain rating of mild, moderate, marked or totally disabled.
* Patients who have undergone total hip arthroplasties in their contralateral hips within the past 12 months.
* Patients with a known allergy to metal (e.g. jewelry).
* Skeletally immature patients (tibial and femoral epiphyses are not closed).
* Evidence of active infections that may spread to other areas of the body (e.g., osteomyelitis, pyogenic infection of the hip joint, overt infection, urinary tract infection, etc.).
* The presence of highly communicable disease or diseases that may limit follow-up (e.g., immuno-compromised conditions, hepatitis, active tuberculosis, etc.).
* Presence of known metastatic or neoplastic disease.
* Significant neurologic or musculoskeletal disorders or disease that may adversely affect gait or weight bearing, (e.g., muscular dystrophy, multiple sclerosis).
* Conditions that may interfere with the total hip arthroplasty's survival or outcome, (e.g., Paget's disease, Charcot's disease).
* Any patient believed to be unwilling or unable to comply with a rehabilitation program for a cementless total hip replacement or who indicates difficulty or inability to return for follow-up visits prescribed by the study protocol.
* Patient is known to be pregnant, a prisoner, mentally incompetent, and/or alcohol or drug abuser.
* Any systemic steroid therapy, excluding inhalers, within three months prior to surgery.
* Patients carrying the diagnosis of inflammatory degenerative arthritis (IDJD) to include the following composite diagnoses: rheumatoid arthritis, systemic lupus erythematosus, pigmented villonodular synovitis, juvenile rheumatory arthritis and other arthritic processes of inflammatory or autoimmune etiology.
* Patients requiring structural bone grafts in order to support the prosthetic component(s) or to shape the bone to receive the implant(s).
* Patients who refuse to provide consent to participate in the clinical investigation.
* Surgical replacement requires the use of an acetabular liner and femoral head greater or smaller than a 36mm diameter

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2003-04-01 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2013-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Politi, MD, Principal Investigator — Cardinal Orthopaedic Institute; Douglas Dennis, MD, Principal Investigator — Colorado Joint Replacement
Locations (5):
- United States (5):
  - Sacramento, California
  - Colorado Joint Replacement, Denver, Colorado
  - Winston-Salem, North Carolina
  - Cardinal Orthopaedic Institute, Columbus, Ohio
  - Alexandria, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected for recruitment into the study from the general diagnosis population defined as "primary total hip arthroplasty (THA) for non-inflammatory degenerative joint disease (NIDJD)." The investigation was conducted at 5 centers. The same inclusion and exclusion criteria applied to both investigational and control groups.
Pre-assignment Details: 1 subject was excluded from the study intraoperatively due to a ceramic liner fracture. Liner fracture was included in the Adverse Event data reported, but the subject was not included in the the number of participants because there are no follow-up data on this subject outside of operative details.
Groups:
- 36 mm Ceramic-on-ceramic: 36 mm ceramic head on ceramic acetabular liner 36 mm ceramic head on a ceramic acetabular liner : Total hip replacement with a 36 mm ceramic head on a ceramic liner
- 28 mm Ceramic-on-polyethylene: 28 mm ceramic-on-polyethylene historical control 28 mm ceramic head on a polyethylene acetabular liner : Total hip replacement with a 28 mm ceramic head on a polyethylene liner.
Period: Overall Study
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Started | 169 | 74
Completed | 150 | 69
Not Completed | 19 | 5

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consists of all enrolled subjects who were implanted with either the investigational or control device. One subject who was randomized to receive the investigational device was exlcuded because of an intra-operative ceramic liner fracture, and hence did not receive the investigational device.
Groups:
- Total: Total of all reporting groups
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene | Total
Number analyzed (Participants) | 168 | 74 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.0) | 56.9 (9.7) | 57.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 27 | 103
  Male | 92 | 47 | 139
Region of Enrollment [Number; unit: participants]
  United States | 168 | 74 | 242

OUTCOME MEASURES:

1. Primary Outcome: Total Harris Hip Score
Description: The Harris Hip scoring system assigns a numeric value to responses from patients and assessments made by a surgeon. A score of 91-100 is excellent, 81-90 is good, 71-80 is fair, 70 or below is poor. The patient records the following: pain level, need for assistance when walking, presence of a limp, distance able to walk, ability to put on shoes and socks, climb stairs, use public transportation and the length of time one is able to comfortably sit in a chair are all scored. The Total Harris Hip Score is a sum of its subscores (Pain, Function, Activities, Deformity, and Range of Motion).
Time Frame: At final follow-up visit, 24 months or later, up to 72 months
Population: The population for this primary endpoint analysis is comprised of subjects who completed the study with a Harris Hip score at final follow-up visit, 24 months or later, through 72 months, minus subjects who were found to have violated a protocol inclusion/exclusion criterion.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 148 | 69
units on a scale | 95.6 (8.8) | 94.9 (8.9)
Statistical Analysis 1: Comparison: 36 mm Ceramic-on-ceramic vs 28 mm Ceramic-on-polyethylene; Test type: Non-Inferiority or Equivalence — The prospectively planned primary endpoint analysis was a non-inferiority test of covariate adjusted 24 month or later Harris Hip score means with a 5 point non-inferiority margin. A prospective power analysis with an anticipated Harris Hip score standard deviation of 10.08 (for both treatment groups) indicated that sample sizes of 134 and 67 would provide approximately 95% statistical power for this non-inferiority test with a type 1 error rate of 5%; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.7, 95% CI 1-sided [lower limit -1.40], Standard Error of Mean 1.24

2. Secondary Outcome: Harris Hip Subscale Score: Pain
Description: The Harris Hip's pain subscale is a numeric value from 0 to 44. A lower score indicates more pain; a score of 44 indicates no pain.
Time Frame: At final follow-up visit, 24 months or later, up to 72 months
Population: The population for this endpoint analysis is comprised of subjects who completed the study with a Harris Hip score at final follow-up visit, 24 months or later, through 72 months, minus subjects who were found to have violated a protocol inclusion/exclusion criterion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 148 | 69
units on a scale | 41.4 (6.3) | 41.1 (5.7)

3. Secondary Outcome: Harris Hip Subscale Score: Function
Description: The Harris Hip's function subscale is a numeric value from 0 to 33. A lower score indicates less function; a score of 33 indicates no limitations in function level.
Time Frame: At final follow-up visit, 24 months or later, up to 72 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 148 | 69
units on a scale | 32.1 (2.5) | 31.6 (4.0)

4. Secondary Outcome: Harris Hip Subscale Score: Activities
Description: The Harris Hip's Activities subscale is a numeric value from 0 to 14. A lower score indicates a lower ability to perform daily activities; a score of 14 indicates no limitations in daily activities.
Time Frame: At final follow-up visit, 24 months or later, up to 72 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 148 | 69
units on a scale | 13.2 (1.4) | 13.0 (1.7)

5. Secondary Outcome: Harris Hip Subscale Score: Deformity
Description: The Harris Hip's Deformity subscale is a numeric value from 0 to 4. A lower score indicates more deformity; a score of 4 indicates no deformity.
Time Frame: At final follow-up visit, 24 months or later, up to 72 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 148 | 69
units on a scale | 4.0 (0) | 4.0 (0)

6. Secondary Outcome: Harris Hip Subscale Score: Range of Motion
Description: The Harris Hip's Range of Motion subscale is a numeric value from 0 to 5. A lower score indicates a lower range of motion; a score of 5 indicates full range of motion.
Time Frame: At final follow-up visit, 24 months or later, up to 72 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 148 | 69
units on a scale | 4.9 (0.1) | 4.9 (0.2)

7. Secondary Outcome: Harris Hip Score Longitudinal Analysis
Description: The Harris Hip scoring system assigns a numeric value to responses from patients and assessments made by a surgeon, with a range of 0 to 100. Lower scores indicate a worse outcome and a score of 100 is the best possible outcome. Longitudinal analysis (repeated measures) was performed to compare post-operative Harris Hip sores over time.
Time Frame: 6 week, 6 month, 12 month, 24 month, 36 month, and 48 months post-operatively
Population: The population for this endpoint analysis is comprised of subjects who had Harris Hip scores at respective follow-up visits minus subjects who were found to have violated a protocol inclusion/exclusion criterion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 148 | 69
units on a scale
  6 week Total Harris Hip Score | 52.6 (10.9) | 52.0 (9.5)
  6 month Total Harris Hip Score | 93.1 (10.0) | 93.4 (9.7)
  12 month Total Harris Hip Score | 95.5 (6.5) | 95.2 (7.6)
  24 month Total Harris Hip Score | 95.7 (8.2) | 93.7 (10.2)
  36 month Total Harris Hip Score | 96.6 (6.8) | 97.0 (4.6)
  48 month Total Harris Hip Score | 94.6 (10.1) | 93.5 (11.1)
Statistical Analysis 1: Comparison: 36 mm Ceramic-on-ceramic vs 28 mm Ceramic-on-polyethylene; A repeated measurements longitudinal model of Harris Hip scores was carried out to compare Harris Hip results between treatment groups across time; Test type: Superiority or Other; p = 0.952, Mixed Models Analysis; SAS PROC MIXED was used with an ante-dependence covariance structure; Mean Difference (Net) = 0.079

8. Secondary Outcome: Proportion of Composite Successes
Description: A subject was deemed to be a composite success at 24 months or greater if at the time of last clinical follow-up there had not been a revision of any THA components, the latest Harris Hip score was 80 or greater, and on the latest radiographic evaluation there were no radiolucencies greater than 2mm, no evidence of acetabular migration greater than 4mm, no change in acetabular shell inclination angle greater than 4 degrees, and no osteolysis.
Time Frame: At final follow-up visit, 24 months or later, up to 72 months
Population: Per Protocol subjects with radiographic endpoints, and including subjects who have been revised (these are composite endpoint failures).
Measure: Number; unit: percentage of participants
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Number analyzed (Participants) | 147 | 71
percentage of participants | 90.5 | 90.1

ADVERSE EVENTS:
Time Frame: Intra-operatively through last follow-up, which was up to 72 months post-op for some subjects.
Description: At study inception, information on whether or not an adverse event was deemed to be serious was not collected. Because of this caveat, the Sponsor has reported all adverse events that occurred in this study
  Note: One (1) subject was excluded from the study intraoperatively due to a ceramic liner fracture. Liner fracture was included in the AE data reported, but was not included in the number of participants because there are no follow-up data on this subject outside of the operative details
Arm/Group | 36 mm Ceramic-on-ceramic | 28 mm Ceramic-on-polyethylene
Serious Adverse Events (participants affected / at risk) | 0/169 | 0/74
Other Adverse Events (participants affected / at risk) | 134/169 | 60/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 36 mm Ceramic-on-ceramic (N=169) | 28 mm Ceramic-on-polyethylene (N=74)
Intra-operative: 2cm non-displaced fracture of posterior femoral neck (Injury, poisoning and procedural complications) | 1/168 | 0
Intraoperative: Blemish on Ceramic Component (General disorders) | 0/168 | 1
Intraoperative: Broken Drill Bit (General disorders) | 1/168 | 0
Intraoperative: Cardiovascular (Cardiac disorders) | 2/168 | 0
Intraoperative: Hematological (Blood and lymphatic system disorders) | 1/168 | 0
Intraoperative: Liner Fracture During Surgery (General disorders) | 1 | 0
Postoperatve Systemic: Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/168 | 3
Postoperative Systemic: Cardiovascular (Cardiac disorders) | 15/168 | 6
Postoperative Systemic: Central Nervous System (Nervous system disorders) | 6/168 | 4
Postoperative Systemic: Dermatological (Skin and subcutaneous tissue disorders) | 8/168 | 0
Postoperative Systemic: Endocrine/Metabolic (Endocrine disorders) | 4/168 | 6
Postoperative Systemic: Gastrointestinal (Gastrointestinal disorders) | 8/168 | 6
Postoperative Systemic: Genitourinary (Renal and urinary disorders) | 10/168 | 7
Postoperative Systemic: HEENT (Ear and labyrinth disorders) | 7/168 | 6
Postoperative Systemic: Hematological (Blood and lymphatic system disorders) | 0/168 | 4
Postoperative Systemic: Musculoskeletal (Musculoskeletal and connective tissue disorders) | 93/168 | 44
Postoperative Systemic: Neurological (Nervous system disorders) | 3/168 | 0
Postoperative Systemic: Other - Fell (Injury, poisoning and procedural complications) | 5/168 | 3
Postoperative Systemic: Other - Insect Bite (Injury, poisoning and procedural complications) | 0/168 | 1
Postoperative Systemic: Pregnancy - 7 Months Gestation (Pregnancy, puerperium and perinatal conditions) | 1/168 | 0
Postoperative Systemic: Peripheral Nervous System (Nervous system disorders) | 4/168 | 3
Postoperative Systemic: Respiratory System (Respiratory, thoracic and mediastinal disorders) | 4/168 | 4
Postoperative Systemic: Thrombosis/Thrombophlebitis (Vascular disorders) | 5/168 | 1
Postoperative Systemic: Wound Problem (Injury, poisoning and procedural complications) | 1/168 | 0
Postoperative Operative Site: Acetabular Component Failure (General disorders) | 1/168 | 0
Postoperative Operative Site: Acetabular Liner Failure (General disorders) | 1/168 | 0
Postoperative Operative Site: Deep Infection (Infections and infestations) | 2/168 | 0
Postoperative Operative Site: Dermatological (Skin and subcutaneous tissue disorders) | 3/168 | 0
Postoperative Operative Site: Dislocation (Injury, poisoning and procedural complications) | 2/168 | 4
Postoperative Operative Site: Femoral Component Loosening (General disorders) | 1/168 | 0
Postoperative Operative Site: Fracture - Femoral Insertional Fx (Injury, poisoning and procedural complications) | 1/168 | 0
Postoperative Operative Site: Hematoma Requiring Drainage (Vascular disorders) | 1/168 | 0
Postoperative Operative Site: Heterotopic Bone Formation (Injury, poisoning and procedural complications) | 3/168 | 0
Postoperative Operative Site: Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4/168 | 0
Postoperative Operative Site: Musculoskeletal (Musculoskeletal and connective tissue disorders) | 16/168 | 3
Postoperative Operative Site: Other - Clicking (Musculoskeletal and connective tissue disorders) | 7/168 | 1
Postoperative Operative Site: Other - Contusion (Injury, poisoning and procedural complications) | 1/168 | 0
Postoperative Operative Site: Other - Fell (Injury, poisoning and procedural complications) | 3/168 | 0
Postoperative Operative Site: Other - Hip Pain (Injury, poisoning and procedural complications) | 2/168 | 1
Postoperative Operative Site: Other - Hip Snapping (Musculoskeletal and connective tissue disorders) | 1/168 | 0
Postoperative Operative Site: Iliopsoas Tendinitis (Musculoskeletal and connective tissue disorders) | 6/168 | 3
Postoperative Operative Site: Other - Squeaking (Musculoskeletal and connective tissue disorders) | 8/168 | 0
Postoperative Operative Site: Other - Stiffness (Musculoskeletal and connective tissue disorders) | 1/168 | 0
Postoperative Operative Site: Subsidence of Femoral Component (General disorders) | 0/168 | 1
Postoperative Operative Site: Other - Vibration (Musculoskeletal and connective tissue disorders) | 1/168 | 0
Postoperative Operative Site: Pain (General disorders) | 8/168 | 2
Postoperative Operative Site: Pain - Thigh (Musculoskeletal and connective tissue disorders) | 6/168 | 3
Postoperative Operative Site: Subluxation (Injury, poisoning and procedural complications) | 1/168 | 0
Postoperative Operative Site: Trochanteric Bursitis (Musculoskeletal and connective tissue disorders) | 17/168 | 4
Postoperative Operative Site: Wound Problem (Injury, poisoning and procedural complications) | 6/168 | 1

LIMITATIONS AND CAVEATS:
At study inception, information on whether or not an adverse event was deemed to be serious was not collected. Because of this caveat, the Sponsor has reported all adverse events that occurred in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less